CLINICAL TRIAL: NCT02323100
Title: A Double Blind, Placebo Controlled, Dose Escalation Trial of Glycerol Phenylbutyrate Corrector Therapy for Cystic Fibrosis
Brief Title: Glycerol Phenylbutyrate Corrector Therapy For CF (Cystic Fibrosis)
Acronym: GPBA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding ended
Sponsor: National Jewish Health (Other)
Collaborators: University of Alabama at Birmingham (Other); Children's Hospital of Philadelphia (Other); Johns Hopkins University (Other); Horizon Pharma Ireland, Ltd., Dublin Ireland (Industry)
Responsible Party: Principal Investigator, Pam Zeitlin, Professor of Pediatrics, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPBA; FD-R-0005380 (Other Grant/Funding Number: FDA Office of Orphan Products Development)
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; corrector; glycerol phenylbutyrate; nasal potential difference
MeSH Terms: conditions — Cystic Fibrosis | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ravicti low dose (Active Comparator): Low dose Ravicti® oral liquid at 6ml (6.6 gm) by mouth or gastrostomy tube at 8 am, 5.5 ml (6.05gm) at 4pm and midnight for 7 days.
  Interventions: Drug: Ravicti low dose
- Ravicti high dose (Active Comparator): Ravicti® oral liquid at 9ml (9.9 gm)at 8 am and 8.25ml (9.08 gm) at 4pm and midnight for 7 days.
  Interventions: Drug: Ravicti high dose
- Placebo (Placebo Comparator): Matching placebo taken at 8am, 4pm and midnight for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ravicti low dose — 8 am, 4pm and midnight
  Other Names: Ravicti, glycerol phenylbutyrate
  Arms: Ravicti low dose
Drug: Ravicti high dose — 8 am, 4pm and midnight
  Other Names: Ravicti, glycerol phenylbutyrate
  Arms: Ravicti high dose
Drug: Placebo — 8 am, 4pm and midnight
  Arms: Placebo

SUMMARY:
We propose to test the effectiveness of the combination of CF pancreatic enzyme replacement therapy (PERT) on absorption of Ravicti® and subsequent restoration of nasal epithelial cystic fibrosis transmembrane conductance regulator (CFTR)-mediated chloride transport during the nasal potential difference (NPD) test. Funding source FDA Office of Orphan Products Development.

DETAILED DESCRIPTION:
We were the first to test 4-phenylbutyrate (Buphenyl) as a systemic corrector of these defects in F508del under an investigator-initiated Investigational New Drug (IND)application held by P. Zeitlin. In a series of Phase 1 and 2 trials we established the maximum tolerated dose as 20 gm daily divided t.i.d. and the maximum induction of cyclic AMP (cAMP)-mediated nasal epithelial chloride transport with 30 gm daily as a median of -10 millivolt (mV) on days 4 and 7 of treatment.1;2 Under those conditions there was no significant decrease in sweat chloride values or in amiloride-inhibited nasal potential difference (NPD). We interpreted these results as a proof of concept of corrector therapy, but corrector therapy alone was likely an insufficient therapy for this mutation in CF, and therefore closed the IND for 4-phenylbutyrate.

In the ensuing years, Vertex Pharmaceuticals, Inc. has had success with the development of ivacaftor3;3;4 (VX-770) as a potentiator of G551D CFTR and has studied the drug alone and in combination with their corrector lumacaftor5 (VX-809) and VX-661. We at Johns Hopkins University (JHU), University of Alabama at Birmingham (UAB) and Childrens' Hospital of Philadelphia/University of Pennsylvania (CHOP/Penn) have participated in many of the clinical trials and are pleased and encouraged by the success of VX-770. It is not yet certain that future combinations of corrector(s) and potentiator(s) will be safe and effective, and it is prudent to explore alternative correctors and potentiators. Furthermore, recent structural investigations in a number of laboratories support the idea that more than one corrector may be necessary to fully restore F508del to the trafficking pathway 6. Precedent for combination of 4PBA with other CFTR modulators has been established in vitro 7;8 4-Phenylbutyrate tablets are formulated for oral delivery, and we showed that the pharmacokinetics were similar in CF to that in patients with urea cycle disorders. However the large number of tablets that had to be ingested at each meal were somewhat daunting at the 30 gm daily dose. A new pro-drug of 4-phenylbutyrate, glycerol phenylbutyrate or Ravicti®(owned by Hyperion Pharmaceuticals, Inc.) was approved in February 2013 by the US FDA. This new formulation is a significant advance for patients with urea cycle disorders because it is an oral, odorless, tasteless liquid, that contains 3 molecules of 4-phenylbutyrate for every molecule of the triglyceride. Simple arithmetic would suggest that one mole equivalent of the pro-drug provides three moles of active drug. However, pancreatic lipase enzymes are required to break the covalent bonds and release the active drug in the intestines. Because most CF patients homozygous for F508del are pancreatic-insufficient and already on enzyme therapy, we propose to test the effectiveness of the combination of CF pancreatic enzyme replacement therapy (PERT) on absorption of Ravicti® and subsequent restoration of nasal epithelial CFTR-mediated chloride transport during the nasal potential difference (NPD) test.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Confirmed diagnosis of CF based on the following criteria:

   any CFTR genotype combination EXCEPT two stop codons, and one or more clinical features consistent with the CF phenotype.
3. Taking pancreatic enzyme replacement therapy (PERT), or have documented pancreatic sufficiency.
4. Ability to perform acceptable spirometry.
5. Ability to understand and sign a written informed consent and comply with the requirements of the study.
6. FEV1 ≥30% of predicted normal for age, gender, and height (Hankinson standards): pre or post-bronchodilator at Screening.
7. Oxygen saturation by pulse oximetry ≥90% breathing either ambient air or regular oxygen regimen at screening and Day 1.
8. Hematology and clinical chemistry of blood and urine results with no clinically significant abnormalities that would interfere with the study assessments (as judged by the principal investigator) at screening. If electrolyte abnormality at screening, values must be corrected prior to dosing.
9. Subjects on chronic inhaled antibiotic therapy are eligible if they can continue their usual antibiotic regimen, or remain on their off-cycle period, for the duration of study drug exposure
10. Negative pregnancy test for women of child-bearing potential.
11. If of childbearing potential, agree to use one highly effective method of contraception from the time of consent through the Visit 4 study visit, per section 9.1.13 of the protocol.

Exclusion Criteria:

1. Administration of any investigational drug or device within 30 days of Screening or within 6 half-lives of the investigational drug (whichever is longer).
2. History of any illness or condition that in the opinion of the investigator could confound the results of the study or pose additional risk in administering study drug to subjects.
3. Any change in chronic therapies for CF lung disease (e.g., Ibuprofen, Pulmozyme®, hypertonic saline, Azithromycin, TOBI®, Cayston®) within 4 weeks of Study Day 1.
4. Pregnant, planned pregnancy or breast feeding at Screening.
5. Clinically significant cardiac, liver or kidney disease.
6. Seizure disorder.
7. Acute upper respiratory infection within 2 weeks or acute pulmonary exacerbation requiring intravenous antibiotics within 4 weeks of Screening Visit.
8. Sinus surgery within 6 weeks of Screening Visit.
9. Abnormal renal function.
10. Abnormal liver function, defined as ≥3x upper limit of normal (ULN), of serum aspartate transaminase (AST) or serum alanine transaminase (ALT), or known cirrhosis.
11. Screening laboratory results which in the judgment of the investigator would interfere with completion of the study.
12. History of or listed for solid organ or hematological transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The primary biological endpoint will be the change in average measurement of nasal potential difference between day 7 and baseline. | 7 days
  chloride and sodium transport in nasal epithelium

SECONDARY OUTCOMES:
Change in other NPD measures from baseline and Days 4, 7, and 14 to include baseline PD, change in amiloride, low chloride, and low chloride plus isoproterenol. | 14 days
  change between date and baseline in sodium and chloride transport
Change in average sweat chloride measurement between days 4, 7, 14 and baseline. | 14 days
  change between study time point and baseline in sweat chloride
Safety and tolerability. | 14 days
  standard safety and tolerability lab values
Efficacy of PERT on absorption of Ravicti®. | 14 days
  quantification of exogenous pancreatic enzyme effects on release of active drug from the pro-drug triglyceride form

OTHER OUTCOMES:
Plasma will be sampled for pharmacokinetics (PK) studies | 14 days
  blood pharmacokinetics
Safety labs: hematology, complete metabolic panel (CMP), C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), uric acid. Sputum microbiology and spirometry will be performed. | 14 days
  blood counts, metabolic measures, CRP

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Zeitlin, MD, PhD, Principal Investigator — National Jewish Health
Locations (3):
- United States (3):
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Johns Hopkins CF research office — http://www.hopkinscf.org/about-us/research-office/